CLINICAL TRIAL: NCT03811561
Title: Long-term Effects of Semaglutide on Diabetic Retinopathy in Subjects With Type 2 Diabetes
Brief Title: A Research Study to Look at How Semaglutide Compared to Placebo Affects Diabetic Eye Disease in People With Type 2 Diabetes
Acronym: FOCUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4352; U1111-1201-6256 (Other: World Health Organization (WHO)); 2017-003619-20 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide once weekly as subcutaneous (s.c., under the skin) injection added to standard of care.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo (semaglutide) once weekly as subcutaneous subcutaneous (s.c., under the skin) injection added to standard of care.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Participants will get one dose of semaglutide once weekly in addition to their diabetes medicines - which treatment they get is decided by chance. Participants will inject the study medicine using a pre-filled PDS290 pen-injector. The medicine must be injected in a skin fold in the stomach, thigh or upper arm once a week. Participants will start with once-weekly doses of 0.25 mg for 4 weeks, then the dose will be gradually increased to 0.5 mg once weekly for 4 weeks, and finally to 1.0 mg once weekly (maximum dose) up to 260 weeks (5 years).
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Participants will get one dose of placebo (semaglutide) once weekly in addition to their diabetes medicines - which treatment they get is decided by chance. Participants will inject the study medicine using a pre-filled PDS290 pen-injector. The medicine must be injected in a skin fold in the stomach, thigh or upper arm once a week. Participants will start with once-weekly doses of 0.25 mg for 4 weeks, then the dose will be gradually increased to 0.5 mg once weekly for 4 weeks, and finally to 1.0 mg once weekly (maximum dose) up to 260 weeks (5 years).
  Arms: Placebo

SUMMARY:
This study will look at the long-term effects of semaglutide (active medicine) on diabetic eye disease when compared to placebo (dummy medicine). The study will be performed in people with type 2 diabetes. Participants will either get semaglutide or placebo in addition to their diabetes medicines - which treatment the participant gets is decided by chance. Participants will inject the study medicine using a pen-injector. The medicine must be injected in a skin fold in the stomach, thigh or upper arm once a week. The study will last for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus.
* HbA1c of 7.0-10.0% (53-86 mmol/mol) (both inclusive).
* Eye inclusion criteria (both eyes must meet all criteria):
* Early Treatment Diabetic Retinopathy Study (ETDRS) level of 10-75 (both inclusive) evaluated by fundus photography and confirmed by central reading centre
* No ocular or intraocular treatment for diabetic retinopathy or diabetic macular oedema six months prior to the day of screening.
* No anticipated need for ocular or intraocular treatment for diabetic retinopathy or diabetic macular oedema within three months after randomisation.
* Best-corrected visual acuity greater than or equal to 30 letters using the ETDRS visual acuity protocol
* No previous treatment with pan-retinal laser photocoagulation
* No substantial non-diabetic ocular condition that, in the opinion of the ophthalmologist, would impact diabetic retinopathy or diabetic macular oedema progression during the trial
* No substantial media opacities that would preclude successful imaging

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within the past 60 days prior to the day of screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of eGFR less than 30 ml/min/1.73 m^2
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods
* Concurrent treatment with any GLP-1 receptor agonist or DPP-4 inhibitor from randomisation.
* Receipt of any investigational medicinal product within 30 days before screening
* Previous participation in this trial. Participation is defined as randomisation
* Known or suspected hypersensitivity to trial products or related products
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-11-07 (Estimated)

PRIMARY OUTCOMES:
Presence of at least 3 steps Early Treatment Diabetic Retinopathy Study (ETDRS) subject level progression. | Year 5
  Percentage of subjects (yes/no).

SECONDARY OUTCOMES:
Time from randomisation to first at least 3 steps ETDRS subject level progression or central involved diabetic macular oedema (ciDME) in either eye. | Up to 5 years
  Measured in months.
Change in visual acuity in the worse seeing eye. | Week 0, Year 5
  Measured in number of letters using the ETDRS protocol.
Change in visual acuity in the better seeing eye. | Week 0, Year 5
  Measured in number of letters using the ETDRS protocol.
Occurrence of treatment for diabetic retinopathy or diabetic macular oedema in either eye with focal/grid laser photocoagulation. | Week 0-Year 5
  Percentage of subjects (yes/no).
Occurrence of treatment for diabetic retinopathy or diabetic macular oedema in either eye with pan-retinal laser photocoagulation. | Week 0-Year 5
  Percentage of subjects (yes/no).
Occurrence of treatment for diabetic retinopathy or diabetic macular oedema in either eye with intravitreal injection with anti-vascular endothelial growth factor (VEGF). | Week 0-Year 5
  Percentage of subjects (yes/no).
Occurrence of treatment for diabetic retinopathy or diabetic macular oedema in either eye with intravitreal injection with steroid. | Week 0-Year 5
  Percentage of subjects (yes/no).
Occurrence of treatment for diabetic retinopathy or diabetic macular oedema in either eye with vitrectomy. | Week 0-Year 5
  Percentage of subjects (yes/no).
Presence of at least 3 steps ETDRS subject level improvement. | Year 5
  Percentage of subjects (yes/no).
Presence of at least 2 steps ETDRS subject level progression. | Year 5
  Percentage of subjects (yes/no).
Presence of at least 2 steps ETDRS subject level improvement. | Year 5
  Percentage of subjects (yes/no).
Presence of persistent visual acuity up to 38 ETDRS letters in either eye. | Year 5
  Percentage of subjects (yes/no).
Presence of persistent at least 2 lines (10 letters) ETDRS worsening in visual acuity in either eye from baseline. | Year 5
  Percentage of subjects (yes/no).
Presence of persistent at least 3 lines (15 letters) ETDRS worsening in visual acuity in either eye from baseline. | Year 5
  Percentage of subjects (yes/no).
Presence of persistent at least 2 lines (10 letters) ETDRS improvement in visual acuity in either eye from baseline. | Year 5
  Percentage of subjects (yes/no).
Persistent at least 3 lines (15 letters) ETDRS improvement in visual acuity in either eye from baseline. | Year 5
  Percentage of subjects (yes/no).
Presence of ciDME in either eye. | Year 5
  Percentage of subjects (yes/no).
Change in glycosylated haemoglobin (HbA1c). | Week 0, Year 5
  Measured in %-points.
Change in body weight. | Week 0, Year 5
  Measured in kg.
Change in systolic and diastolic blood pressure. | Week 0, Year 5
  Measured in mmHg.
Change in Lipids: Total-cholesterol, High density lipoprotein (HDL)-cholesterol, low density lipoprotein (LDL)-cholesterol and triglycerides. | Week 0, Year 5
  Measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (226):
- United States (72):
  - Synexus Rsch /Cnt Phnx Med C, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - South Arizona VA Healthcare System, Tucson, Arizona
  - Synexus Cln Rsrch Inc - Orange Gro FP, Tucson, Arizona
  - Southern California Res Ctr, Coronado, California
  - FDRC, Costa Mesa, California
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Diabetes/Lipid Mgmt & Res Ctr, Huntington Beach, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Angel City Research, Inc., Los Angeles, California
  - Downtown LA Res Ctr. Inc., Los Angeles, California
  - Riverside University Health System Medical Center, Moreno Valley, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Clinical Trials Research_Sacramento_0, Sacramento, California
  - UCLA Diabetes Center at Santa Monica, Santa Monica, California
  - Coastal Metabolic Research Center, Ventura, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Rocky Mount Reg VA Med-DN, Aurora, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Innovative Research of W FL, Clearwater, Florida
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - Apex Medical Research Inc, Chicago, Illinois
  - The University Of Chicago, Chicago, Illinois
  - American Health Network of Indiana, LLC_Avon, Avon, Indiana
  - American Health Network of Indiana, LLC_Greenfield, Greenfield, Indiana
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - VA Medical Center, Lexington, Kentucky
  - Kentucky Diabetes-Endocrinology Center, Lexington, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston Medical Center_Cary, Boston, Massachusetts
  - Joslin Center For Diabetes, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Synexus Clinical Research US, Inc._Tempe_0, Richfield, Minnesota
  - Diabetes & Endo Specialists Inc, Chesterfield, Missouri
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern New Hampshire Diabete, Nashua, New Hampshire
  - Lovelace Scientific Resources Inc, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - NYC Research, Inc., New York, New York
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Harold Hamm Diabetes Center, Oklahoma City, Oklahoma
  - Aria Endocrine Metabolic Assoc, Philadelphia, Pennsylvania
  - Tristar Clin Investigations, PC, Philadelphia, Pennsylvania
  - Holston Medical Group Pc, Bristol, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Vanderbilt Diab Obes Clin Tri, Nashville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Synexus Clinical Research US, INC., Murray, Utah
  - MultiCare Inst for Res & Innov, Spokane, Washington
- CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo, Brazil
- Bulgaria (12):
  - DCC I- Pleven EOOD Endocrinology, Pleven
  - MHAT Sveti Pantaleimon - Pleven, Internal Diseases, Pleven
  - MHAT Med Line Clinic, Plovdiv
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Endocrinology, Plovdiv
  - MHAT MC-Sv Ivan Rilski EOOD, Plovdiv
  - "DCC VII - Sofia", Endocrinology Consulting Room, Sofia
  - DCC VII - Sofia EOOD, Endocrinology, Sofia
  - MHAT Knyaginya Klementina - Sofia EAD, Sofia
  - USHATE Akad. Ivan Penchev EAD, Second Clinic of Endocrinology, Sofia
  - IV MHAT - Sofia EAD, Sofia
  - DCC XX - Sofia EOOD, Endocrinology, Sofia
  - Medical centre Vitclinic EOOD, Sofia
- Canada (9):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - LMC Clinical Res Thornhill, Concord, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - LMC Oakville, Oakville, Ontario
  - The Ottawa Hospital_Riverside, Ottawa, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - LMC Clinical Research, Inc. (Montreal Glen), Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Diabetologie Krupska, Prague
  - Fakultni nemocnice Kralovske Vinohrady_Praha, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - MUDr. Michala Pelikanova, Prague
- Germany (9):
  - Praxis Denger/Pfitzner, Friedrichsthal, Friedrichsthal
  - Diabetologische Schwerpunktpraxis Harburg- Dr. med.Paschen,, Hamburg
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Wendisch - Dahl Hamburg - DZHW, Hamburg
  - Wendisch/Dahl Hamburg, Hamburg
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
- Greece (7):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - Iatriko Psychicou Private Clinic, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - University Hospital of Athens ATTIKON, Haidari-Athens
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
- India (25):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Narayana Hrudayalya Institute of Cardiac Sciences, Bangalore, Karnataka
  - Diacon Hospital Private Limited, Bangalore, Karnataka
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Indian Institute of Diabetes, Thiruvananthapuram, Kerala
  - Indian Institute of Diabetes, Thiruvnanthapuram, Kerala
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Government Medical College and Super Speciality Hospital, Nagpur, Nagpur, Maharashtra
  - DEW Medicare & Trinity hospital, Nagpur, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, Ansari Nagar, New Delhi 110029, New Delhi
  - Apollo Hospital, Delhi, New Delhi
  - Indraprastha Apollo Hospital, Delhi, New Delhi
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Dayanand Medical College & Hospital_Ludhiana, Ludhiana, Punjab
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Arthur Asirvatham hospital,, Madurai, Tamil Nadu
  - SSKM, Kolkata, West Bengal
  - Apollo Gleneagles Hospital, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Care Hospital, Hyderabad
  - Aditya Jyot Hospital, Mumbai
- Israel (6):
  - Rambam MC - Diabetes and obesity center of excellence, Haifa
  - Hadassah Ein Karam MC - Diabetes Unit, Jerusalem
  - Meir MC - Diabetes unit, Kfar Saba
  - Rabin MC Beilinson - Endo unit, Petah Tikva
  - Sourasky MC - Institute of Endocrinology, metabolism and hypertension, Tel Aviv
  - Sheba MC - Endocrinology Clinic, Tel Litwinsky
- Latvia (5):
  - Zemgales diabetes centre, Jelgava
  - Teterovska practice, Ogre
  - P. Stradins Clinical University Hospital, Riga
  - Medical Centre Pulss 5, Riga
  - Juglas Medicine Center, Riga
- Mexico (2):
  - Instituto Nacional de Nutricion - Unidad de Inv de Enf Metab, Distrito Federal, México, D.F.
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
- Poland (16):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - In-Vivo Sp. z o.o., Bydgoszcz
  - B_Serwis Popenda Sp.J., Chorzów
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - NZOZ Gdanska Poradnia Cukrzycowa Sp.z o.o., Gdansk
  - Centrum Medyczne Pratia Katowice, Katowice
  - Clinical Medical Research Korfantego - Ambulatoryjna Opieka, Katowice
  - FutureMeds Sp. z o.o., Krakow
  - Santa Sp. z o.o, Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - Prywatny Gabinet Lekarski Jan Ruxer, Lodz
  - NZOZ "DiabMed" Poradnia Diabetologiczna, Poznan
  - Gaja Poradnie Lekarskie, Poznan
  - SPZZOZ im. Marszalka J. Pilsudskiego w Plonsku, Płońsk
  - SPSK nr 1 im. prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, ul. 3-go Maja 13/15 41-800 Zabrze, Zabrze
  - Santa Sp. z o.o, Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz, Łódź Voivodeship
- Portugal (9):
  - ULS De Matosinhos E.P.E.- Hospital Pedro Hispano, Senhora Da Hora, Matosinhos, Matosinhos
  - ULS Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - ULS Da Regiao De Aveiro E.P.E. - Hospital Infante D. Pedro, Aveiro
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - ULS Do Alto Ave, E.P.E. - Hospital Senhora da Oliveira - Guimarães, Guimarães
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Centro Hospitalar de São João, Porto
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - ULS Da Arrábida, E.P.E._Hospital de São Bernardo, Setúbal
- Romania (7):
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Clinic of Diabetes Cluj, Cluj-Napoca, Cluj
  - SC Centru Medical Dr. Negrisanu SRL, Timișoara, Timiș County
  - 3rd Clinic for Nutrition-Spitalulul Județean de Urgenta, Timișoara, Timiș County
  - "Carol Davila" Military Emergency Hospital, Bucharest
  - Sana Monitoring SRL, Bucharest
  - SC Clinica Diabnutrimed S.R.L., Bucharest
- Russia (14):
  - Multispecialty Medical Clinic Anturium LLC, Barnaul
  - Kazan Federal University, Kazan'
  - PIH "Clin Hosp "RZD-Medicina" former Kazan OJSC Rus Railways, Kazan'
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - National Medical Research Center of Endocrinology, Moscow
  - Branch of limited liability company "Hadassah Medical LTD", Moscow
  - State Novosibirsk regional clinical hospital, Novosibirsk
  - City Consultative & Diagnostic Centre #1, Saint Petersburg
  - Diagnistic Centre "Energo", Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Llc "International Medical Center "Time", Saint-Peterburg
  - SHI Saratov City Clinical Hospital #9, Saratov
  - Regional clinical cardiology dispensary, Saratov
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Serbia (5):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Centre Nis, Endocrinology, Diabetes and Metabolism, Niš
- Slovakia (5):
  - V. interna klinika LF UK a UNB, Bratislava
  - Nemocnica akademika L. Derera, UNB, Bratislava
  - Diabetologicka ambulancia, Dia Zilina s.r.o., Žilina
  - Medivasa s.r.o., Diabetologicka ambulancia, Žilina
  - MEDIVASA, s.r.o., Diabetologicka ambulancia, Žilina
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Virgen de la Macarena, Seville
  - Hospital La Fe - Endocrinología y Nutrición, Valencia
- United Kingdom (10):
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Queen's Medical Centre University Hospital, Nottingham, Nottinghamshire
  - University Hospital, Queens Medical Centre, Nottingham, Nottinghamshire
  - Yeovil District Hospital - Clinical Research Unit, Yeovil, Somerset
  - Kings College Hospital, London
  - Norfolk and Norwich University Hospital, Norfolk
  - George Eliot Hospital NHS Trust, Nuneaton
  - George Eliot Hospital, Nuneaton
  - Clinical Research Unit, Somerset
  - Royal Cornwall Hospital (Treliske), Truro

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com